CLINICAL TRIAL: NCT03606083
Title: Prospective Multicenter Registry to Examine the Real-world Performance of the E-liac Stent Graft System for Treatment of Uni- or Bilateral Aorto-iliac or Iliac Aneurysms
Brief Title: Registry in Patients With Aorto-iliac or Iliac Aneurysms
Acronym: PLIANTII
Status: Active, not recruiting | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PLIANTII
Record Dates: First submitted 2018-06-29; First posted 2018-07-30 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Vascular Aneurysm
Keywords: aorto-iliac; iliac; aneurysm
MeSH Terms: conditions — Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular repair — Endovascular repair of aorto-iliac or iliac aneurysms using an iliac branch device (IBD)

SUMMARY:
The PLIANT II registry is undertaken to examine the real-world outcome after treatment of consecutive patients with uni- or bilateral aorto-iliac or iliac aneurysms using the E-liac Stent Graft System.

DETAILED DESCRIPTION:
In this study, patients will be observed who receive one or two E-liac Stent Graft(s) for aorto-iliac or iliac aneurysms. The E-liac Stent Graft(s) will be implanted at the discretion of the treating physician. Participating physicians will be asked to provide their observations collected during routine care for patients he/she had decided to treat with the E-liac Stent Graft System. Informed consent of the patients to allow the use of their clinical records for the purpose of this observational study will be obtained before intervention and before data are being collected.

The period of data collection will be 60 months starting from the intervention for each patient. 100% verification of patient informed consent and essential study documents will be performed at each study site. 60% of patient´s source documentation will be randomly monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Patient must have an aorto-iliac or iliac aneurysm
* Patient must have a unilateral or bilateral iliac aneurysm
* Patient´s anatomy must be suitable for stent graft placement on preoperative angio CT scan
* Patient must be available for the appropriate follow-up times for the duration of the study
* Patient has been informed of the nature of the study, agrees to its provisions and has signed the informed consent form prior to intervention

Exclusion Criteria:

* Female of child bearing potential
* Patients with ruptured iliac aneurysms
* Patients with juxtarenal, pararenal or suprarenal aneurysms
* Patients pretreated with Nellix (Endologix) or Altura (Lombard Medical)
* Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints
* Patient with malignancy needing chemotherapy or radiation
* Patients with life expectancy of less than 3 years
* Patient minor or under guardianship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with uni- or bilateral aorto-iliac or iliac aneurysm, treated with the E-liac Stent Graft System.
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from endoleak type I or III and patency of EIA and IIA on E-liac implantation side(s) | 12 months
  Rate of patients that reach the primary endpoint

SECONDARY OUTCOMES:
Mortality | 24 hours
  Rate of all cause mortality in peri-operative periods
Survival rate | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of survival
Aneurysm size | 12, 24, 36, 60 months
  Rate of patients with decreasing, stable, increasing aneurysm size
Primary patency of EIA / IIA | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with primary patency of EIA / IIA
Secondary patency of EIA / IIA | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with secondary patency of EIA / IIA
Stent graft dislodgement | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with stent graft dislodgement
Endoleak type I | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with infrarenal type Ia endoleak
Endoleak type Ia in the CIA (isolated iliac aneurysm treatment) | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with infrarenal type Ia endoleak
Endoleak type Ib in the CIA | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with endoleak type Ib in the CIA
Endoleak type Ib in the EIA | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with endoleak type Ib in the EIA
Endoleak type Ib in the IIA | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with endoleak type Ib in the IIA
Endoleak type II | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with endoleak type II
Endoleak type III | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with endoleak type III
Stent fracture | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with stent fracture
Reintervention | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate patients with reintervention after E-liac Stent Graft implantation
Claudication | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with increasing, stable, decreasing claudication (walking distance without pain)
Adverse Events | prior to discharge / 30 days, 12, 24, 36, 60 months
  Rate of patients with adverse events (product-related, procedure-related, aneurysm-related)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brunkwall, Prof., Principal Investigator — Cologne University Hospital
Locations (1):
- Universitätsklinikum Köln, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anton S, Wiedner M, Stahlberg E, Jacob F, Barkhausen J, Goltz JP. Initial Experience with the E-liac(R) Iliac Branch Device for the Endovascular Aortic Repair of Aorto-iliac Aneurysm. Cardiovasc Intervent Radiol. 2018 May;41(5):683-691. doi: 10.1007/s00270-017-1868-x. Epub 2018 Jan 3. PMID 29299625
- [Background] Mylonas SN, Rumenapf G, Schelzig H, Heckenkamp J, Youssef M, Schafer JP, Ahmad W, Brunkwall JS; E-liac Collaborative Group. A multicenter 12-month experience with a new iliac side-branched device for revascularization of hypogastric arteries. J Vasc Surg. 2016 Dec;64(6):1652-1659.e1. doi: 10.1016/j.jvs.2016.04.065. Epub 2016 Aug 1. PMID 27492764
- [Result] Oberhuber A, Deglise S, Richter O, Makaloski V, Bracale U, Isernia G, Tines R, Cappelli A, Dorweiler B, Brunkwall J; PLIANTII Study Collaboration. A Prospective, Multicentre Registry on Thirty Day and One Year Outcomes of the E-liac Stent Graft System in Patients with Unilateral or Bilateral Aorto-iliac or Iliac Aneurysms: The PLIANTII Study. Eur J Vasc Endovasc Surg. 2025 Jun;69(6):847-854. doi: 10.1016/j.ejvs.2025.02.029. Epub 2025 Feb 20. PMID 39986435